CLINICAL TRIAL: NCT04393467
Title: Efficacy of Transcranial Static Magnetic Field Stimulation (tSMS) in Amyotrophic Lateral Sclerosis (ALS).
Brief Title: Transcranial Static Magnetic Field Stimulation (tSMS) in Amyotrophic Lateral Sclerosis (ALS).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Full Professor of Neurology, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STIMALS
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; transcranial magnetic stimulation; static magnetic field; tSMS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tSMS (Experimental): tSMS will be delivered by a magnet applied to M1, bilaterally (120 min daily, for 6 months). Magnet will be kept in position by a plastic helmet.
  Interventions: Device: tSMS
- sham tSMS (Sham Comparator): A non-magnetic steel cylinder, with same size, weight and appearance of the magnet, will be used for sham stimulation.
  Interventions: Device: sham tSMS

INTERVENTIONS:
Device: tSMS — tSMS delivered on bilateral motor cortex
  Arms: real tSMS
Device: sham tSMS — sham tSMS delivered on bilateral motor cortex by a non-magnetic steel cylinder, with same size, weight and appearance of the magnet used for real tSMS
  Arms: sham tSMS

SUMMARY:
This study aims to evaluate safety and efficacy of tSMS in ALS patients and to obtain preliminary data about the effects of tSMS on cortical excitability.

To this purpose, 40 ALS patients will be recruited and randomized to real or sham tSMS. After at least 3 months follow-up, they will undergo tSMS, daily for 120 min, at home, for 6 consecutive months.

Clinical status will be tested before, during and after the stimulation period. Moreover, cortical excitability will be tested by transcranial magnetic stimulation (TMS) before and after the stimulation period.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* diagnosis of ALS according to revised El Escorial criteria and Awaji-Shima criteria
* disease duration < 24 months
* ALSFRS-R > 30 at the recruitment
* ALSFRS-R decline > 1 in the at least 3-months period before the intervention
* normal respiratory functionality (FVC > 80% and ALSFRS-R items 10,11,12 > 4) at the recruitment
* treatment with riluzole 50 mg x 2/die

Exclusion Criteria:

* inclusion in other clinical trials
* presence of tracheotomy or/and PEG (percutaneous endoscopic gastrostomy)
* contraindications to magnetic fields exposure
* pregnancy or breast-feeding
* history of epilepsy or seizures
* assumption of drugs acting on central nervous system, except for antidepressive drugs and benzodiazepines.
* cognitive impairment
* lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 9 months
  Comparison between the ALSFRS-R (Revised Amyotrophic Lateral Sclerosis Functional Rating Scale) decline over the period of at least three months before the treatment and the period of six months during the treatment. The ALSFRS-R is 12-items scale ranking from 0 (worse) to 48 (better) points.

SECONDARY OUTCOMES:
Safety and tolerability | 6 months
  Incidence of adverse events during the stimulation period
Compliance | 6 months
  Number of stimulation sessions actually completed by each patient
Effect on resting motor threshold (RMT) and active motor threshold (AMT) | 6 months
  Change in TMS-derived cortical excitability parameters (RMT and AMT) before and after stimulation period.
Effect on motor evoked potentials (MEP) size | 6 months
  Change in TMS-derived cortical excitability parameters (MEP size) before and after stimulation period.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Neurology and Laboratory of Neuroscience, Istituto Auxologico Italiano, IRCCS, Milan
  - Neurology Unit, Campus Biomedico University, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Lazzaro V, Ranieri F, Doretti A, Boscarino M, Maderna L, Colombo E, Soranna D, Zambon A, Ticozzi N, Musumeci G, Capone F, Silani V. Transcranial static magnetic stimulation for amyotrophic lateral sclerosis: a bicentric, randomised, double-blind placebo-controlled phase 2 trial. Lancet Reg Health Eur. 2024 Jul 30;45:101019. doi: 10.1016/j.lanepe.2024.101019. eCollection 2024 Oct. PMID 39185360